CLINICAL TRIAL: NCT06197685
Title: A Novel Combinatory Approach to Maximize Functional Recovery of Learning and Memory in Multiple Sclerosis
Acronym: COMBINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Carly Wender, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R123323
Record Dates: First submitted 2023-12-04; First posted 2024-01-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Aerobic exercise; Virtual Reality; Leg cycling; Mobility disability
MeSH Terms: conditions — Multiple Sclerosis | interventions — beta-Aminoethyl Isothiourea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the intent of the two exercise conditions. The outcomes assessor will also be blinded to the random assignment of enrolled participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Rehabilitation + Aerobic Exercise with Virtual Reality (VR) (Experimental): In the cognitive rehabilitation and aerobic exercise with VR condition, participants will complete a supervised, aerobic exercise training program (AET) integrated with virtual reality (Ideally Designed Exercise to Accelerate Learning/memory; IDEAL) three days per week over a 12 week period. For seven weeks, participants will only complete IDEAL. For weeks 8-12, participants will complete the Kessler Foundation modified story Memory Technique (KF-mSMT®), a memory retraining program on 2 of the 3 days per week.
  Interventions: Behavioral: The Kessler Foundation modified Story Memory Technique® (KF-mSMT®); Behavioral: Aerobic Exercise Training (AET) plus Virtual Reality (IDEAL)
- Cognitive Rehabilitation + Stretching and Toning (Experimental): In the cognitive rehabilitation and stretching and toning (S/T) exercise condition, participants will complete 12 weeks of supervised S/T activities 3 days per week over the 12 week period. For seven weeks, participants will only complete S/T. During weeks 8-12, participants will complete the Kessler Foundation modified story Memory Technique (KF-mSMT®), a memory retraining program on 2 of the 3 days per week.
  Interventions: Behavioral: The Kessler Foundation modified Story Memory Technique® (KF-mSMT®); Behavioral: Stretching and Toning (S/T)

INTERVENTIONS:
Behavioral: The Kessler Foundation modified Story Memory Technique® (KF-mSMT®) — KF-mSMT is a memory retraining technique that consists of two-related skills: (1) imagery and (2) context/organization. The proposed KF-mSMT intervention includes 10 total sessions with 2 sessions per week for 5 weeks. Each session will last 45-60 minutes.
Behavioral: Aerobic Exercise Training (AET) plus Virtual Reality (IDEAL) — The AET condition includes 12 weeks of supervised, progressive, moderate intensity cycle ergometry. The AET will include semi-immersive, interactive VR such the cycling speed on the bike will translate directly to perceived speed through the virtual environment.
  Other Names: IDEAL
  Arms: Cognitive Rehabilitation + Aerobic Exercise with Virtual Reality (VR)
Behavioral: Stretching and Toning (S/T) — The S/T condition will include 12 weeks of supervised S/T activities that target the head/neck. shoulder, elbow/forearm, hand/wrist, trunk/hip, ankle/foot.
  Arms: Cognitive Rehabilitation + Stretching and Toning

SUMMARY:
The goal of this novel study is to compare the effect of a combined cognitive rehabilitation and exercise approach on new learning and memory (NLM) in persons with multiple sclerosis (pwMS) and mobility disability.

DETAILED DESCRIPTION:
The proposed research study will be the first to apply the Kessler Foundation modified Story Memory Technique (KF-mSMT®), the practice standard for cognitive rehabilitation, with one of two exercise programs. Alone, KF-mSMT® has been beneficial to NLM impairment, however, its effects are highly selective to list learning and as such, will not maximally restore NLM function. The combination of KF-mSMT® and exercise provides a robust approach towards maximal functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Be within the ages of 18 and 70 years of age
* Speak English as their primary language
* Confirmed MS diagnosis by a neurologist
* Be relapse and steroid-free for at least 30 days
* Mild-to-moderate self-reported mobility disability, based on the Patient Determined Disease Steps scale (PDDS)
* Currently physically inactive, based on the Godin Leisure Time Exercise Questionnaire (GLTEQ)
* Right handedness

Exclusion Criteria:

* History of neurological disorders besides MS or history of uncontrolled psychiatric disorders (ex: major depression)
* Have contraindications to exercise, based on the Physical Activity Readiness Questionnaire (PAR-Q)
* Currently use medications that may impact cognition (ex: steroids, benzodiazepines)
* Currently pregnant
* Contraindication for MRI (metal or electronic devices in the body that are not considered MRI safe)
* Severe cognitive impairment as measured by the Modified Telephone Interview of Cognitive Status (TICS-M)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in objective new learning and memory (NLM). | Weeks 1 and 2 (pre-intervention) and Weeks 15 and 16 (post-intervention)
  The California Verbal Learning Test-Second Edition (CVLT-II) measures verbal learning and memory by having participants recall a list of words from 4 semantic categories. The word list is presented over 5 trials with a 20 minute delayed recall and recognition trial. Standardized T-scores range from 0-100, where higher scores indicated better performance.
Change in everyday memory | Weeks 1 and 2 (pre-intervention) and Weeks 15 and 16 (post-intervention)
  The Ecological Memory Simulations (EMS) is a multi-component test that measures memory as it relates to everyday life. Scores range from 0-205, where higher scores indicated better performance.

SECONDARY OUTCOMES:
Change in hippocampal volume | Weeks 1 and 2 (pre-intervention) and Weeks 15 and 16 (post-intervention)
  MRI data will be collected in the Rocco Ortenzio Neuroimaging Center at Kessler Foundation using an FDA-approved 3.0 T Siemens Skyra scanner and a 32-channel head coil to measure the volume of bilateral hippocampi.
Change in hippocampal function | Weeks 1 and 2 (pre-intervention) and Weeks 15 and 16 (post-intervention)
  fMRI data will be collected during a list-learning task conducted while in the FDA-approved 3.0 T Siemens Skyra scanner with a 32-channel head coil.

CONTACTS AND LOCATIONS:
Overall Officials: Carly Wender, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No